CLINICAL TRIAL: NCT02300844
Title: Investigation on Safety, Tolerability and Pharmacokinetics of Single Doses of NNC0174-0833 in Normal Weight, Overweight to Obese But Otherwise Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9838-3993; U1111-1131-7160 (Other: WHO)
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC0174-0833 10 mg/mL (Experimental)
  Interventions: Drug: NNC0174-0833
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0174-0833 — Subjects will receive a single s.c. (subcutaneous/under the skin) dose of NNC0174-0833.
  Up to nine dose levels of single s.c. doses of NNC0174-0833 are planned to be investigated.
  Arms: NNC0174-0833 10 mg/mL
Drug: placebo — Subjects will receive a single s.c. (subcutaneousl/under the skin) dose.
  Arms: Placebo

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to investigate the safety, tolerability and pharmacokinetics of single doses of NNC0174-0833 in normal weight, overweight to obese but otherwise healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight, Overweight or obese (Body Mass Index [BMI]) between or equal to 20.0 and 35.0 kg/m^2 but otherwise healthy men
* Age between or equal to 22 and 64 years at the time of signing informed consent

Exclusion Criteria:

* History of, or presence of, cancer, diabetes or any clinically significant cardiovascular,respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders including sleep apnoea, as judged by the investigator
* Subjects with history of, or presence of, a disease being associated with impaired calcium homeostasis and/or increased bone turnover (e.g. Paget´s disease, osteoporosis)
* Male subjects of reproductive age who are not using a highly effective physical barrier method of contraception (sexual abstinence, or condom with spermicidal foam/gel/film/cream) combined with a method with Pearl Index less than 1% for their nonpregnant partner(s) (such as implants, injectables, combined oral contraceptives, hormonal intrauterine devices or diaphragm+spermicide, or surgical sterilisation or post-menopausal) and/or who intend to donate sperm in the period from start of Visit 2 up to 3 months following the administration of the investigational medicinal product

Ages: 22 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From the time of dosing (Day 1) until completion of the post treatment follow-up visit (Day 43-50)

SECONDARY OUTCOMES:
Area under the NNC0174-0833 plasma concentration-time curve | Prior to the initial dose on day 1 and 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 48, 60, 72, 96, 120, 168, 240, 336, 504, and 1008 hours post-dose
Maximum concentration of NNC0174-0833 in plasma | Prior to the initial dose on day 1 and 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 48, 60, 72, 96, 120, 168, 240, 336, 504, and 1008 hours post-dose
Time to maximum concentration of NNC0174-0833 in plasma | Prior to the initial dose on day 1 and 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 48, 60, 72, 96, 120, 168, 240, 336, 504, and 1008 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com